CLINICAL TRIAL: NCT02829580
Title: Evaluation of Non-invasive Endothelial Function in Children Sickle by Vascular Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 07 307 02; 07 307 02 (Other: Local grant)
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Sickle Cell Disease
Keywords: endothelial function; flow-mediated dilation; vascular elastic properties
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sickle group (Experimental): Children with major sickle cell syndrome will have an usual Echocardiography
  Interventions: Procedure: Echocardiography
- Control group (Active Comparator): Children recruited in a previous study and who had an usual Echocardiography
  Interventions: Procedure: Echocardiography

INTERVENTIONS:
Procedure: Echocardiography — Measures by Doppler and study of endothelial function

SUMMARY:
Sickle cell disease (SCD) is an inherited disorder characterized by recurrent painful crises with ischemia resulting from vascular occlusion. Adults with SCD have increased arterial stiffness and reduced flow-mediated dilation (FMD), due to impaired release of substances such as nitric oxide.

The present study assess the vascular properties of carotid and brachial arteries in children with SCD compared with a control group without cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

Sickle cell group :

* Children with sickle cell syndrome (SS or SC)
* Children hospitalized in the hematology unit (day hospital)
* The girls set must have had a negative pregnancy test.
* One of the two holders of parental authority must have signed consent form
* Children affiliated to a social security scheme or equivalent

Control group : Children recruited in a previous study :

* Holders of parental authority affiliated to a social security scheme
* Children recruited during the balance of a heart murmur or a vasovagal reaction
* Children whose cardiological examination is normal
* Children having no cardiovascular risk factor

Exclusion Criteria:

Sickle cell group :

* Children with intercurrent diseases such as obesity, intra uterine growth retardation (IUGR), hypertension, renal failure, infectious diseases (including HIV, Hepatitis C) or chronic inflammatory
* Children who have sickle cell crisis there is less than 1 month.

Control group :

Children with intercurrent diseases: obesity, IUGR, hypertension, renal failure, infectious diseases (including HIV, Hepatitis C) or chronic inflammatory

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2008-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of endothelial function | baseline
  Evaluation parameter of endothelial function (brachial artery): flow dependent dilatation (expressed in%)

SECONDARY OUTCOMES:
match the measurement thickness of the intima media | baseline
  The thickness of the intima media (ITM) on the right common carotid
match the measurement systolic and diastolic diameters | baseline
  systolic and diastolic diameters (sD, dD)
distensibility cross sectional | baseline
  match the measurement on the compliance and distensibility cross sectional (CCS, DCS)
Match the measurement on the diastolic wall stress | baseline
  diastolic wall stress (DWS)

CONTACTS AND LOCATIONS:
Overall Officials: DULAC YVES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hadeed K, Hascoet S, Castex MP, Munzer C, Acar P, Dulac Y. Endothelial Function and Vascular Properties in Children with Sickle Cell Disease. Echocardiography. 2015 Aug;32(8):1285-90. doi: 10.1111/echo.12851. Epub 2014 Dec 3. PMID 25470331